CLINICAL TRIAL: NCT07240727
Title: An Investigation of the Effects of Different Practical Roles in Simulation-Based Intermediate Life Support Training on Theoretical Knowledge, Practical Skill Acquisition, and Self-Assessment Among Undergraduate Dental Students
Brief Title: The Effect of Role Differences on Learning and Self-Assessment in Simulation-Based Life Support Training Among Dental Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gözde Nur Erkan (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Sponsor-Investigator, Gözde Nur Erkan, Assisstant Professor, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KU-ERKAN-005
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Intermediate Life Support; Dental Students; Self Evaluation; Peer Assessment; Instructor Guidance; OSCE (Objective Structured Clinical Examination)
Keywords: Intermediate Life Support (ILS); Dental Education; Simulation-based Training; Self-assessment; Peer Assessment; Instructor Assessment; OSCE

STUDY DESIGN:
Intervention Model Description: All participants receive the same intermediate life support (ILS) educational program. After the initial theoretical and practical training, students are divided into two groups: one group assumes the practitioner role in simulation-based practical sessions, while the other group serves as evaluators. Both groups participate in observations and assessments, including self-assessment, peer assessment, and instructor assessment. No experimental intervention is applied; the study measures the development of theoretical knowledge and practical skills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Practitioner
  Interventions: Other: Intermediate Life Support (ILS) Educational Program: Practitioner
- Group 2 (Active Comparator): Evaluator
  Interventions: Other: Intermediate Life Support (ILS) Educational Program-Evaluator

INTERVENTIONS:
Other: Intermediate Life Support (ILS) Educational Program: Practitioner — Students assigned to the practitioner arm participate in simulation-based practical sessions, taking the active role in managing adult, pediatric, and infant cardiac and respiratory arrest scenarios. They perform all steps of intermediate life support (ILS), including detection of arrest, chest compressions, positive-pressure ventilation with 100% oxygen, calling emergency services (112), and requesting emergency equipment. Practitioner students may act as single or multiple rescuers during simulations, and each student assumes a leadership role at least once.
  Arms: Group 1
Other: Intermediate Life Support (ILS) Educational Program-Evaluator — Students assigned to the evaluator arm observe practitioner students during simulation-based practical sessions. They use checklists based on current AHA and ERC guidelines to assess the practitioners' performance and provide immediate feedback. Evaluators also complete self-assessment to measure their own perception of knowledge and practical skills.
  Arms: Group 2

SUMMARY:
This study aims to evaluate the effectiveness of theoretical and practical training on intermediate life support (ILS) among fifth-year dental students. Participants will be assigned to two roles during simulation-based sessions: practitioners, who perform the interventions, and evaluators, who assess peers using structured checklists. The study will compare theoretical knowledge and practical skills before and after the training, and assess the impact of peer evaluation on learning outcomes. A minimum of 84 students will be enrolled to ensure adequate statistical power. The results will inform the optimization of dental education in emergency life support training.

DETAILED DESCRIPTION:
This study aims to investigate the development of theoretical knowledge and practical skills of fifth-year dental students through pre- and post-training assessments, and to compare outcomes between study groups. Prior to receiving theoretical instruction, students will complete a baseline knowledge questionnaire to assess their initial theoretical understanding. Similarly, an initial practical assessment using an Objective Structured Clinical Examination (OSCE) will be conducted to determine baseline practical competence.

Following detailed theoretical training and practical exercises, students will be divided into two groups for simulation-based practical sessions:

Group 1 (Practitioners): Students in this group will participate as practitioners in additional practical sessions following joint theoretical and practical training.

Group 2 (Evaluators): Students in this group will serve as evaluators during the additional practical sessions, using structured checklists developed with the instructor.

During the ILS simulation exercises, practitioner students are expected to detect cardiac and respiratory arrest in adult and pediatric scenarios and implement acute management steps, including activating emergency services (calling 112), requesting an automated external defibrillator, and utilizing emergency intervention equipment. Practitioners will perform chest compressions and positive pressure ventilation with 100% oxygen using appropriate devices. To simulate single- or multi-rescuer interventions, practitioner students will perform in groups of one or two, while evaluators observe and provide immediate feedback. Each student will assume a leadership role at least once, with assisting students following the leader's instructions.

Evaluator students will assess practitioner performance using checklists aligned with the latest American Heart Association (AHA) and European Resuscitation Council (ERC) Basic and Advanced Life Support guidelines. Evaluators will provide immediate feedback on any deficiencies or errors. After simulation sessions, students will undergo OSCE assessments encompassing both adult and pediatric scenarios to evaluate practical skills and theoretical knowledge acquisition. Assessments will be conducted by instructors using rubrics and checklists based on current AHA and ERC recommendations. In addition, students will perform self-assessments using the same rubrics to evaluate their own perception of competence. A minimum of 20 teams will be evaluated three times throughout the study: by the instructor, by their peers, and through self-assessment, enabling the monitoring of skill development and self-evaluation accuracy over time.

Inclusion Criteria:

Fifth-year students enrolled in the Faculty of Dentistry.

Exclusion Criteria:

Students unwilling to participate.

Students with more than 10% absenteeism in training sessions where missed content cannot be made up.

ELIGIBILITY:
Inclusion Criteria:

* Fifth-year students currently enrolled in the Faculty of Dentistry.

Exclusion Criteria:

* Students who declined to participate in the study were excluded.
* Students who demonstrated more than 10% absenteeism from the training sessions, where the missed sessions could not be made up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in theoretical knowledge and practical skill scores across two time points during Intermediate Life Support (ILS) training | Baseline (pre-training) and Post-training (within 20 minutes during pre and post training OSCE sessions)
  Theoretical knowledge and practical skill levels of fifth-year dental students will be evaluated using written tests and Objective Structured Clinical Examinations (OSCEs) administered at two time points: before the training (baseline) and after the completion of the training (post-training). Changes in scores across these time points will be analyzed to assess learning and clinical skill competence progression.

SECONDARY OUTCOMES:
Change and accuracy of self-assessment scores compared with peer and instructor evaluations during Intermediate Life Support (ILS) training | After each of the three simulation sessions (Session 1, Session 2, Session 3) (within 10 minutes during each sessions)
  Evaluator and practitioner students will complete self-assessment rubrics after each of three simulation-based practical sessions. These self-assessments will be conducted for a minimum of 20 student teams. Scores will be compared with corresponding peer and instructor evaluations to assess the development and accuracy of students' self-assessment abilities over time. The analysis will evaluate both intra-individual improvement and agreement with external assessments across the three evaluation rounds.
Quality of written documentation and feedback provided by students during the final OSCE | At the final OSCE (post-training assessment), (within 15 minutes during third OSCE station)
  During the final OSCE (Objective Structured Clinical Examination), students will complete a written documentation task describing their approach to the simulated case and provide open-ended as well as rubric-based feedback regarding the training process.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Faculty of Dentistry, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data generated in this study will be made available by the corresponding author upon reasonable request